CLINICAL TRIAL: NCT04940429
Title: Oculometric Assessment of Dynamic Visual Processing in Patients With Obesity and the Impact of Bariatric Surgery
Brief Title: Eye Movement Testing in Patients With Obesity and the Impact of Weight Loss Surgery
Status: Terminated | Type: Observational
Why Stopped: collaboration with research partner stopped, Covid
Sponsor: Stanford University (Other)
Collaborators: Neurofit Inc, Mountain View, California (Unknown)
Responsible Party: Principal Investigator, POkafor, Clinical Assistant Professor, Stanford University
Other Study IDs: 45650
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid
Keywords: Oculometrics
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Roux n Y Gastric Bypass (RYGB): Participants in this arm will include patients who will be having a RYGB after their assessment by their bariatric surgeon. After reviewing and signing the consent form, participants will perform the paper-based standard psychometric tests (number connection test A and B, line tracing test, and digital subtraction test, and serial dotting test, which take about 20 minutes) at their preoperative visit.
  After completion of paper-based standard psychometric tests, participants will then perform the computer application test which takes about 5 minutes at their preoperative visit.
  These will also be performed at their post operative visits 2 weeks, 3, 6 and 12 months.
  Interventions: Device: Neurofit; Diagnostic Test: Psychometric hepatic encephalopathy score
- Sleeve gastrectomy (SG): Participants in this arm will include patients who will be having a SG after their assessment by their bariatric surgeon. After reviewing and signing the consent form, participants will perform the paper-based standard psychometric tests (number connection test A and B, line tracing test, and digital subtraction test, and serial dotting test, which take about 20 minutes) at their preoperative visit.
  After completion of paper-based standard psychometric tests, participants will then perform the computer application test which takes about 5 minutes at their preoperative visit:
  These will also be performed at their post operative visits 2 weeks, 3, 6 and 12 months.
  Interventions: Device: Neurofit; Diagnostic Test: Psychometric hepatic encephalopathy score

INTERVENTIONS:
Device: Neurofit — This involves sitting on a chair with a head and chin rest to maintain stability. Patients will then follow a moving object on the computer screen with their eyes which allows estimation of individual oculometrics along with a composite score. No physical contact or placement of invasive devices will be performed.
Diagnostic Test: Psychometric hepatic encephalopathy score — During the number connection tests, the participant is asked to join dots between numbers or numbers and letters in a timed fashion and the number of seconds required is the outcome. In the line tracing test, participants are required to trace a line between two parallel lines and the time required is noted. Also, the number of times the subject strays outside the line (line tracing test error) is captured. In the digit symbol test, participants are required to pair numbers with special symbols. An individual's score reflects the number of correct pairs achieved in 120 seconds. In the serial dotting test, participants are asked to dot the center of a group of blank circles and the time required to complete the test is the outcome. Psychometric tests will be completed at their post-operative visits.

SUMMARY:
Obesity is a condition of chronic low-grade inflammation, thought to be secondary to adipose tissue secretion of cytokines including interleukin 6 (IL-6), and tumor necrosis factor alpha (TNF- α) which effect multiple pathways and lead to an increase in C-reactive protein (CRP), a sensitive marker of systemic inflammation. Chronic inflammation is thought to be a major risk factor for the development of metabolic syndrome, diabetes, cardiovascular disease and cancer. Inflammatory cytokines have also been shown to directly and indirectly interact with the central nervous system influencing behavior and neural activity.

Obesity is an independent risk factor for reduced cognitive function including poor attention, executive function and memory. Demonstrating improvement in dynamic visual processing following bariatric surgery could expand our understanding of the impact of obesity on central nervous system (CNS) function.

DETAILED DESCRIPTION:
This study will involve the utilization of a noninvasive computer application (Neurofit) to perform oculometric assessment of dynamic visual processing . Eye movements are short latency, voluntary motor behaviors that consist of various aspects including visual motion, pursuit initiation, steady-state tracking, direction tuning, and speed tuning. The computer application is based on an eye movement methodology that can quantify many aspects of human dynamic visual processing using a noninvasive video-based eye tracking technology with validated oculometric analysis techniques. It captures 8 domains of oculometric function and reports a composite score (NFit).

Prior studies have demonstrated sensorimotor dysfunction in patients with diffuse brain injury which leads to derangement in information processing throughout the brain. This computer application has been utilized in patients with traumatic brain injury (TBI). Liston et al, in a study of 34 TBI patients, demonstrated that TBI patients had several individual oculometrics that were significantly deranged including pursuit latency, initial pursuit acceleration, pursuit gain, catch-up saccade amplitude, proportion smooth tracking, and speed responsiveness.

By comparing individual and composite oculometric data between patients before and after weight-loss surgery, this research study hopes to identify any significant differences or distinct patterns that may exist as a result of obesity. We also intend to compare changes in high-sensitivity CRP to assess if post-surgical changes in this inflammatory marker correlates with improvement in dynamic visual processing. Patients seen in our bariatric surgery clinic are primarily offered Roux-en-Y gastric bypass (RYGB) and sleeve gastrectomy (SG) as surgical weight loss options. These two procedures are different in that while both provide significant weight loss, the hormonal effects are different between procedures. For this reason, patients undergoing both surgeries will be recruited to determine any differences in oculometrics and serum biomarkers by surgery type. Liver histology data will be obtained per chart review if previously available. This data will be used to ascertain the existence of fatty liver disease, steatohepatitis and/or cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are overweight or obese (Body Mass Index over 25 and 30, respectively)

Exclusion Criteria:

* Individuals <18 years
* Patients with history of cognitive brain disease including traumatic brain injury, dementia, Parkinson's disease
* Individuals with uncontrolled neuropsychiatric illnesses or overt hepatic encephalopathy
* Ongoing alcohol or illicit substance use
* patients with cirrhosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients being considered for weight loss surgery by their bariatric surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Nfit score | Baseline to 1 year post operatively
  Composite oculometric testing score on Neurofit

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No